CLINICAL TRIAL: NCT03170505
Title: Using of Acellular Dermal Matrix in Cleft Palatal Fistula and Compare With Use of Conchal Cartolage
Status: Completed | Type: Observational
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Meisam AbdarEsfahani, Using of Acellular Dermal Matrix in cleft palatal fistula and compare with Use of Conchal Cartolage, Isfahan University of Medical Sciences
Other Study IDs: 29750
Record Dates: First submitted 2017-05-26; First posted 2017-05-31 (Actual); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Cleft Palate
Keywords: cleft palate
MeSH Terms: conditions — Cleft Palate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Acellular Dermal Matrix
  Interventions: Procedure: repairing fistula
- Conchal Cartilage
  Interventions: Procedure: repairing fistula

INTERVENTIONS:
Procedure: repairing fistula — A tailored piece of Acellular Dermal Matrix or Conchal Cartilage will be placed between the oral and nasal layers for repair of a Cleft Palate.

SUMMARY:
The fact that still exist is which method for repairing of secondary cleft palatal fistula is the best. This study will have shown whether using of Acellular dermal Matrix decreased the fistula formation versus using Conchal Cartilage during secondary fistula. Among studies that published, they have not consensus for using acellular dermal matrix. Most of the questions are about cost effectiveness, time that surgery and rehabilitation need and patient risk ( risk of transmission disease from other human tissue )

DETAILED DESCRIPTION:
Observational study composed of a prospective cohort group receiving ADM compared to a retrospective historical cohort group with Conchal Cartilage.

Primary objectives:

The primary objective of this study is to determine whether ADM would lower the incidence of palatal fistula in patients undergoing secondary cleft palate fistula repair.

Secondary objectives:

1. hypo nasality speech after surgery
2. Improvement Speech Score

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed as having cleft palate fistula, with ADM will be included in this study.

Exclusion Criteria:

* Selection will be based on the patient's willingness to allow to participate in the study.
* Patients with diagnosed craniofacial syndromes will be excluded from the study.
* Children with known wound healing defects, will be excluded from the study.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients who present to the Isfahan Cleft palate Clinic with a cleft palate fistula that undergo surgical repair
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2015-05-27 (Actual); Primary Completion 2017-05-27 (Actual); Study Completion 2017-05-27 (Actual)

PRIMARY OUTCOMES:
Fistula formation | Within 2 year of surgery